CLINICAL TRIAL: NCT02476825
Title: A Randomized, Open-labelled Bronchoscopy Study to Assess the Effects of Inhaled Corticosteroids (ICS) on Adult Healthy Volunteers
Brief Title: A Bronchoscopy Study to Assess the Effects of Inhaled Corticosteroids on Adult Healthy Volunteers
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospitals, Leicester (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 168769
Record Dates: First submitted 2015-06-17; First posted 2015-06-19 (Estimated); Last update posted 2023-12-06 (Actual); Status verified 2023-05

CONDITIONS: Healthy
Keywords: volunteers
MeSH Terms: interventions — Fluticasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Inhaled fluticasone (Active Comparator): Inhaled fluticasone propionate (via dry powder inhaler [Accuhaler]), 500 micrograms b.i.d. for 4 weeks
  Interventions: Drug: Fluticasone propionate; Device: Accuhaler
- Observational (No Intervention): Observation

INTERVENTIONS:
Drug: Fluticasone propionate — Flixotide Accuhaler 500 micrograms b.i.d.
  Other Names: Flixotide
  Arms: Inhaled fluticasone
Device: Accuhaler — Flixotide Accuhaler 500 micrograms b.i.d.
  Arms: Inhaled fluticasone

SUMMARY:
This is a randomized, single-blind, controlled, single centre bronchoscopy study designed to assess the effects of fluticasone propionate on airway gene expression and cellularity in healthy adult controls without asthma.

DETAILED DESCRIPTION:
This is a randomized, single-blind, controlled, single centre bronchoscopy study designed to assess the effects of fluticasone propionate on airway gene expression and cellularity in healthy adult controls without asthma. This study will allow a more accurate assessment of the changes in gene/protein expression and cellularity that drive severe treatment-resistant asthma by allowing for the effects that are due to corticosteroids rather than the disease to be considered. This improved mechanistic understanding is important to identify novel therapeutic targets in severe asthma, and to support the development of novel therapeutics. The primary endpoint is the corticosteroid-inducible gene expression pattern in healthy airways.

Approximately 30 healthy adult subjects (age 18-65) will be randomised in a 2:1 ratio to one of two study groups: i) patients will receive fluticasone propionate 500 mcg b.i.d. via Accuhaler for 4 weeks (n=20), or ii) patients will receive no treatment for 4 weeks (n=10). Bronchoscopy will be performed in all patients at baseline, prior to the start of the treatment period and at the end of week 4. The PI, Genentech and Leicester laboratory support staff will be blinded to treatment allocation. A control arm is included to assess the repeatability of the planned analyses, the stability of the gene expression profiles measured during this study period, and to provide a comparator to the treatment group.

Written informed consent for participation in the study must be obtained before performing any study-specific tests or evaluations. Consent will be obtained at the screening visit. At screening, important co-morbidities will excluded . Patients will also be randomised at this screening visit.

To ensure there are sufficient data for analysis, if a subject withdraws before completion of the study, they will be replaced with another subject.

ELIGIBILITY:
Inclusion Criteria:

* Participant willing and able to give informed consent
* Male or Female, aged 18-65 years at Visit 1
* Forced expiratory volume at one second (FEV1) >80% predicted
* FEV1/forced vital capacity (FVC) ratio ≥70%
* Non-smoker for >1 year with <10 py smoking history
* Female participants of child bearing potential must ensure use of effective contraception during the study
* Participants has clinically acceptable laboratory and ECG at screening
* A chest x-ray confirming the absence of significant lung disease
* A negative result to skin prick testing with common aeroallergens, or, if a skin prick test to a common aeroallergen is positive, a negative response to challenge with methacholine (defined as a provocative concentration causing a 20% fall in FEV1 [PC20 methacholine] >16 mg/ml)
* Able (in the Investigators opinion) and willing to comply with all study requirements

Exclusion Criteria:

* Failure to meet the inclusion criteria
* Female participants who are pregnant, lactating or planning pregnancy during the course of the study
* History of a severe allergic reaction or anaphylaxis to corticosteroids
* Systemic treatment with corticosteroids within last 6 months
* Any infection that resulted in hospital admission for ≥ 24 hours within 4 weeks prior to Visit 1 or during screening
* Any infection that required treatment with IV or intramuscular (IM) antibiotics within 4 weeks prior to Visit 1 or during screening
* Any active infection that required treatment with oral antibiotics within 2 weeks prior to Visit 1 or during screening
* Upper or lower respiratory tract infection within 4 weeks prior to Visit 1 or during screening
* Active tuberculosis requiring treatment within 12 months prior to Visit 1
* Known immunodeficiency including but not limited to HIV infection
* Evidence of acute or chronic hepatitis or known liver cirrhosis
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT), or total bilirubin elevation ≥2.0 × the upper limit of normal (ULN) during screening
* Clinically significant abnormality on screening ECG or laboratory tests (haematology, serum chemistry, and urinalysis) that, in the opinion of the investigator, may pose an additional risk in administering study drug to the patient or performing bronchoscopy
* Known current malignancy or current evaluation for a potential malignancy
* Unable to safely undergo elective flexible fiberoptic bronchoscopy because of any one of the following:
* History of allergic reaction to local anesthetics to be used during the bronchoscopy
* Presence of clinically significant abnormality on Screening Coagulation Panel
* Presence of clinically significant medical comorbidities that, in the opinion of the investigator, may make the patient unsuitable for elective bronchoscopy or would impact on study efficacy assessments
* A history of atopic disease (allergic rhinitis [perennial or seasonal], atopic dermatitis, food allergy)
* History of alcohol or drug abuse that would impair or risk the patient's full participation in the study, in the opinion of the investigator
* Current smoker, former smoker with smoking history of >10 pack-years.
* Treatment with anticoagulant medications including but not limited to aspirin,warfarin or antiplatelet medication
* Use of a licensed or investigational monoclonal antibody within 6 months or 5 drug half-lives prior to Visit 1 (whichever is longer)
* Use of a systemic immunomodulatory or immunosuppressive therapy within 6 months or 5 drug half-lives prior to Visit 1 (whichever is longer).
* Use of other investigational therapy not described above within 6 months or 5 drug half-lives prior to Visit 1 (whichever is longer)
* Receipt of a live attenuated vaccine within 4 weeks prior to Visit 1
* Use of complementary, alternative, or homeopathic medicines including, but not limited to traditional or non-traditional herbal medications within 3 months
* Scheduled elective surgery or other procedures requiring general anaesthesia during the study
* Donation of blood during the study or within the past 12 weeks
* BMI >38 kg/m2
* Body weight <40 kg

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-01-20 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Relative change from baseline in airway tissue gene expression following 4-weeks of inhaled fluticasone propionate treatment | 6 months after last patient visit

SECONDARY OUTCOMES:
Relative change from baseline in airway cellularity following 4-weeks of inhaled fluticasone propionate treatment | 18 months after last patient visit
Relative change from baseline in airway protein expression following 4-weeks of inhaled fluticasone propionate treatment | 18 months after last patient visit
Relative change from baseline in peripheral blood gene expression following 4-weeks of inhaled fluticasone propionate treatment | 18 months after last patient visit
Differentiate pathways, biomarkers, and heterogeneity between gene expression and pathophysiology in severe asthmatics on ICS +/- lebrikizumab (separate Genentech-sponsored study known as CLAVIER) and healthy volunteers on ICS | 18 months after last patient visit

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bradding, DM, Principal Investigator — University of Leicester/University Hospitals of Leicester NHS Trust
Locations (1):
- University Hospitals of Leicester NHS Trust, Leicester, Leics, United Kingdom

REFERENCES:
- [Derived] Marchi E, Hinks TSC, Richardson M, Khalfaoui L, Symon FA, Rajasekar P, Clifford R, Hargadon B, Austin CD, MacIsaac JL, Kobor MS, Siddiqui S, Mar JS, Arron JR, Choy DF, Bradding P. The effects of inhaled corticosteroids on healthy airways. Allergy. 2024 Jul;79(7):1831-1843. doi: 10.1111/all.16146. Epub 2024 Apr 30. PMID 38686450